CLINICAL TRIAL: NCT05411809
Title: The ctDNA for Evaluating Whether to Use Adjuvant Therapy After SBRT in Patients With Early Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-SBRT
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Stereotactic Body Radiation Therapy
MeSH Terms: interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1 (No Intervention): The ctDNA is positive after SBRT and no adjuvant therapy is used after SBRT.
- Arm 2 (Experimental): The ctDNA is positive after SBRT and adjuvant therapy is used after SBRT.
  Interventions: Drug: drug adjuvant therapy
- Arm 3 (No Intervention): The ctDNA is negative after SBRT and no adjuvant therapy is used after SBRT.

INTERVENTIONS:
Drug: drug adjuvant therapy — The adjuvant treatment regimens depend on the judgment of oncology physicians according to pathological type, molecular characteristics and other details of the tumor.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether ctDNA could help to evaluate whether to use drug adjuvant therapy after SBRT in patients with early lung cancer.

DETAILED DESCRIPTION:
This is a prospective study. The purpose of this study is to determine whether MRD could help to evaluate whether to use drug adjuvant therapy after SBRT in patients with early lung cancer. The ctDNA was detected for early stage lung cancer patients before and after SBRT. If a high level of ctDNA was detected after SBRT, the patients were randomly divided into observation group and adjuvant treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed as non-small cell lung cancer, and was early stage（AJCC 8th）;
2. Patients aged between 18 -80 years; with expected survival time>3 months.
3. Patients with normal organ function within 30 days prior to treatment, the following criteria are met:

   1. blood routine examination criteria : i) hemoglobin (HB) ≥90g/L; ii) absolute neutrophil count (ANC) ≥1.5×10e9/L; iii) platelet (PLT) ≥80×10e9/L; b) biochemical tests meet the following criteria: i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN; iii) serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr) ≥60mL/min;

Exclusion Criteria:

1. Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer);
2. Patients with factors that affect oral medication (such as cannot swallow, chronic diarrhea and intestinal obstruction, etc.) or intravenous medication;
3. Patients with any other severe and/or uncontrolled disease;
4. Patients with a history of psychotropic medicine abuse and cannot quit or have mental disorders;
5. Patients with disease which will severely endanger their security and could not complete this study, according to the judgement of researchers；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
PFS | 3-year
  progression-free survival

SECONDARY OUTCOMES:
PFS | 5-year
  progression-free survival
OS | 3-year
  overall survival
OS | 5-year
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology Cancer Center, Peking University Third Hospital 49# North Garden Rd.,Haidian Dist., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No